CLINICAL TRIAL: NCT02542215
Title: A Multicenter, Randomized, Placebo-controlled, Double-blinded Study of the Efficacy, Safety, and Pharmacokinetics of Cobiprostone for the Prevention of Severe Oral Mucositis in Subjects With Head and Neck Cancer (HNC)
Brief Title: Cobiprostone for the Prevention of Oral Mucositis in Subjects With Head and Neck Cancer Receiving Concurrent Radiation and Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCMP-8811-202
Record Dates: First submitted 2015-08-13; First posted 2015-09-04 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2016-08

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis | interventions — cobiprostone; Drug Therapy; Radiation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cobiprostone 30 mcg four times daily (Experimental): Cobiprostone oral spray, four times daily, in addition to standard care radiation and chemotherapy
  Interventions: Drug: Cobiprostone; Drug: Standard Care - Chemotherapy; Radiation: Standard Care - Radiation
- Placebo 0 mcg four times daily (Placebo Comparator): Matching placebo oral spray, four times daily, in addition to standard care radiation and chemotherapy
  Interventions: Drug: Placebo; Drug: Standard Care - Chemotherapy; Radiation: Standard Care - Radiation

INTERVENTIONS:
Drug: Cobiprostone — Cobiprostone 30 mcg oral spray
  Other Names: SPI-8811
  Arms: Cobiprostone 30 mcg four times daily
Drug: Placebo — Matching placebo oral spray
  Other Names: Placebo comparator
  Arms: Placebo 0 mcg four times daily
Drug: Standard Care - Chemotherapy — Chemotherapy, as given with radiation as standard care for patients with head and neck cancer.
  Other Names: Chemotherapy
Radiation: Standard Care - Radiation — Radiation, as given with chemotherapy as standard care for patients with head and neck cancer.
  Other Names: Radiation

SUMMARY:
Treatment for head and neck cancer often involves a combination of chemotherapy and radiation.

One of the unfortunate consequences of standard care for head and neck cancer is the development of painful mouth sores, known as oral mucositis.

This study will evaluate the use of cobiprostone spray to prevent oral mucositis, when given for the duration of radiation and chemotherapy (RT/CT) standard care.

ELIGIBILITY:
Inclusion Criteria:

* Recently-diagnosed (within the last 6 months), histologically-documented, non-metastatic squamous cell carcinoma of the oral cavity and/or oropharynx amenable to radiotherapy with concurrent chemotherapy as the definitive treatment modality.
* Clinical treatment plan calls for a minimum of 50 Gy cumulative radiation dose administered via continuous course of external beam irradiation to the oral cavity and/or oropharynx via intensity-modulated radiation therapy (IMRT) and/or image-guided radiation therapy (IGRT), combined with conventional or weekly/tri-weekly cisplatin or carboplatin chemotherapy regimen.

Exclusion Criteria:

* Subject has received prior radiation to the head and neck region (+/- chemotherapy).
* Subject has had any other prior invasive malignancy, unless disease-free for a minimum of 3 years.
* Subject has metastatic disease (M1) Stage IV-C.
* Subject has a presence of mucosal ulceration or oral mucositis at screening or develops this prior to randomization, and/or has unhealed wounds remaining from surgical resection and/or excisional biopsy procedure.
* Subject is using a pre-existing feeding tube for nutritional support at study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a diagnosis of severe oral mucositis during the course of receiving up to 50 Gray (Gy) cumulative radiation dose administration with concurrent chemotherapy | 50 Gray (Gy), up to 12 weeks
Overall mean Area Under the Curve (AUC) of oral mucositis severity over time | 50 Gray (Gy), up to 12 weeks

SECONDARY OUTCOMES:
Time-to-onset of severe [World Health Organization (WHO) grade 3 or 4] oral mucositis following initiation of RT/CT | 50 Gray (Gy), up to 12 weeks
Duration of severe (World Health Organization [WHO] grade 3 or 4) oral mucositis | 50 Gray (Gy), up to 12 weeks
Weekly Quality of Life assessment [MD Anderson Symptom Inventory Head and Neck Cancer Module (MDASI-HN)] | 50 Gray (Gy), up to 12 weeks
Mean cumulative radiation dose at time of severe (WHO grade 3 or 4) oral mucositis onset | 50 Gray (Gy), up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (75):
- United States (75):
  - Investigational Site, Birmingham, Alabama
  - Investigational Site, Peoria, Arizona
  - Investigational Site, Yuma, Arizona
  - Investigational Site, Little Rock, Arkansas
  - Investigational Site, Duarte, California
  - Investigational Site, Fullerton, California
  - Investigational Site, Los Angeles, California
  - Investigational Site, Montebello, California
  - Investigational Site, Oceanside, California
  - Investigational Site, Redondo Beach, California
  - Investigational Site, San Francisco, California
  - Investigational Site, Whittier, California
  - Investigational Site, Denver, Colorado
  - Investigational Site, Farmington, Connecticut
  - Investigational Site, Fort Lauderdale, Florida
  - Investigational Site, Fort Myers, Florida
  - Investigational Site, Lakeland, Florida
  - Investigational Site, Miami Beach, Florida
  - Investigational Site, Naples, Florida
  - Investigational Site, Plantation, Florida
  - Investigational Site, Stuart, Florida
  - Investigational Site, Winter Haven, Florida
  - Investigational Site, Boise, Idaho
  - Investigational Site, Urbana, Illinois
  - Investigational Site, Fort Wayne, Indiana
  - Investigational Site, South Bend, Indiana
  - Investigational Site, Topeka, Kansas
  - Investigational Site, Ashland, Kentucky
  - Investigational Site, Baton Rouge, Louisiana
  - Investigational Site, Metairie, Louisiana
  - Investigational Site, New Orleans, Louisiana
  - Investigational Site, Shreveport, Louisiana
  - Investigational Site, Baltimore, Maryland
  - Investigational Site, Bethesda, Maryland
  - Investigational Site, Burlington, Massachusetts
  - Investigational Site, Ann Arbor, Michigan
  - Investigational Site, Detroit, Michigan
  - Investigational Site, East Lansing, Michigan
  - Investigational Site, Minneapolis, Minnesota
  - Investigational Site, St Louis, Missouri
  - Investigational Site, Billings, Montana
  - Investigational Site, Omaha, Nebraska
  - Investigational Site, Reno, Nevada
  - Investigational Site, Egg Harbor, New Jersey
  - Investigational Site, New Brunswick, New Jersey
  - Investigational Site, Charlotte, North Carolina
  - Investigational Site, Gastonia, North Carolina
  - Investigational Site, Greenville, North Carolina
  - Investigational Site, Canton, Ohio
  - Investigational Site, Sylvania, Ohio
  - Investigational Site, Oklahoma City, Oklahoma
  - Investigational Site, Coos Bay, Oregon
  - Investigational Site, Corvallis, Oregon
  - Investigational Site, Portland, Oregon
  - Investigational Site, Gettysburg, Pennsylvania
  - Investigational Site, Hershey, Pennsylvania
  - Investigational Site, Natrona Heights, Pennsylvania
  - Investigational Site, Philadelphia, Pennsylvania
  - Investigational Site, Pittsburgh, Pennsylvania
  - Investigational Site, State College, Pennsylvania
  - Investigational Site, Pawtucket, Rhode Island
  - Investigational Site, Myrtle Beach, South Carolina
  - Investigational Site, Cookeville, Tennessee
  - Investigational Site, Austin, Texas
  - Investigational Site, Fort Sam Houston, Texas
  - Investigational Site, Galveston, Texas
  - Investigational Site, Houston, Texas
  - Investigational Site, Temple, Texas
  - Investigational Site, Charlottesville, Virginia
  - Investigational Site, Fort Belvoir, Virginia
  - Investigational Site, Bellingham, Washington
  - Investigational Site, Everett, Washington
  - Investigational Site, Seattle, Washington
  - Investigational Site, Morgantown, West Virginia
  - Investigational Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No